CLINICAL TRIAL: NCT06346743
Title: Comparison of Effects of Fenofibrate Adjuvant Therapy Versus Conventional Phototherapy in Treatment of Neonatal Exaggerated Hyperbilirubinemia.
Brief Title: Comparison of Effects of Fenofibrate Adjuvant Therapy Versus Conventional Phototherapy in Neonatal Jaundice.
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Muhammad Zark (Other Government)
Responsible Party: Sponsor-Investigator, Muhammad Zark, Postgraduate Resident, Services Institute of Medical Sciences, Pakistan
Organization: Services Institute of Medical Sciences, Pakistan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB/2023/1119/SIMS
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Physiological Neonatal Jaundice; Physiological Hyperbilirubinaemia
Keywords: Phototherapy; Fenofibrate; Hyperbilirubinaemia; Neonatal Jaundice; Fenofibrate Adjuvant Phototherapy
MeSH Terms: conditions — Jaundice, Neonatal; Hyperbilirubinemia | interventions — Fenofibrate; Phototherapy

STUDY DESIGN:
Intervention Model Description: To compare the effects of Fenofibrate adjuvant to phototherapy with conventional phototherapy for exaggerated neonatal hyperbilirubinemia in the form of bilirubin reduction, duration of phototherapy, hospital stay & observation of side-effects.
  After informed consent, single dose of Fenofibrate will be given to the group A (intervention group) and Group B (non-intervention) will only be given phototherapy. Then every 24-hourly sample for serum bilirubin will be sent for lab analysis, for 3 days. A randomized control trial is conducted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fenofibrate adjuvant therapy (Experimental): Single dose fenofibrate adjuvant to conventional phototherapy
  Interventions: Drug: Fenofibrate; Device: Phototherapy
- Conventional phototherapy (Active Comparator): Only conventional phototherapy
  Interventions: Device: Phototherapy

INTERVENTIONS:
Drug: Fenofibrate — Single dose of Fenofibrate will be given at dose of 10mg/Kg along with phototherapy for 24 hours before next blood sampling
  Other Names: Fenofibrate adjuvant phototerapy
  Arms: Fenofibrate adjuvant therapy
Device: Phototherapy — only phototherapy will be given for 24 hours before next blood sampling
  Other Names: conventional bluelight phototherapy

SUMMARY:
Neonatal jaundice has significant importance in neonatal morbidity and mortality world-wide. Though phototherapy has a relentless use in neonatal jaundice, its cumbersome side effects and the physical separation of baby from the mother eventually result as increase in days of hospitalization adding to the mental anguish of the parents. This study is conducted to observe the reduction of serum bilirubin level in neonates treated with Fenofibrate as an adjuvant to phototherapy in treatment of exaggerated physiological hyperbilirubinemia. After informed consent, single dose of Fenofibrate will be given to the group A (intervention group) and Group B (non-intervention) will only be given phototherapy. Then every 24-hourly sample for serum bilirubin will be sent for lab analysis, for 3 days. A randomized control trial is conducted and later on, the data will be analyzed in the SPSS 26. Quantitative variables like age will be presented as mean ± SD. Qualitative variables like gender will be presented as percentage and frequency. Comparison of two groups intervention group and non-intervention group, apply independent sample t-test. P value < 0.05 will be taken as significant. Limitation of the proposed study includes limited sample size, study population limited to only one hospital and no follow-up in plan. If the role of Fenofibrate is established in the management of exaggerated physiological hyperbilirubinemia in newborns, it will be beneficial to minimize the risk of the complications, rapid regression of hyperbilirubinemia & shortening the length of hospital stay.

DETAILED DESCRIPTION:
Neonatal jaundice has significant importance in neonatal morbidity and mortality worldwide. Bilirubin is an antioxidant against the free radical which is circulating in neonatal biological system. Elevation in the serum bilirubin levels readily manifest as jaundice in newborns and this could be attributed to the physiological immaturity of the hepato-biliary system in the neonates. Apart from this increased bilirubin production, less effective binding and transportation, inefficient conjugation and excretion and increased entero-hepatic circulation make a newborn vulnerable for hyperbilirubinemia (Prabha et al., 2020).

Various studies have shown that risk factors for hyperbilirubinemia include low birth weight, breastfeeding, neonatal infection, premature rupture of membrane, male gender, East Asian race, and bleeding during the first trimester of pregnancy. Indirect hyperbilirubinemia is dangerous and can cause kernicterus. ABO and Rh incompatibility, sepsis, breast milk, hypothyroidism, deficiency of a particular enzyme (e.g., glucose-6-phosphate dehydrogenase [G6PD], Gilbert's syndrome, and hypertrophic pyloric stenosis cause indirect hyperbilirubinemia (Watchko et al., 2018).

Management of neonatal jaundice includes identification of neonates at risk, evaluating the underlying cause of pathological hyperbilirubinemia, deciding the thresholds for initiating and stopping treatment and following up of neonates with severe hyperbilirubinemia. Phototherapy remains as the principal modality of treatment in treating severe hyperbilirubinemia where light of blue green spectrum with the wavelength corresponding with peak absorption by bilirubin (450-460nm) is used. Though phototherapy has a relentless use in neonatal jaundice, its cumbersome side effects and the physical separation of baby from the mother eventually result as increase in days of hospitalization adding to the mental anguish of the parents (Prabha et al., 2020).

The pharmacological treatment now under trial for hyperbilirubinemia are metalloporphyrins, penicillamine, phenobarbitate, zinc sulfate and fibrates. Fibrates induces bilirubin conjugation much more readily and effectively. It converts unconjugated bilirubin to conjugated bilirubin thereby hasten its clearance. Fenofibrate as an adjuvant to phototherapy in term neonate with pathological jaundice is well tolerated and associated with significant reduction of serum bilirubin levels, a shorter duration of phototherapy, shorter hospital stay and higher frequency of exclusive breast-feeding, without significant adverse effects in either the single or double dosage. (Awad et al., 2020) In a systemic review, the results of the five studies showed the significant effect of Fenofibrate as adjuvant therapy on reducing TSB level, the meta-analysis failed to show the same result in the study groups. (Zamiri et al., 2020) Fenofibrate as an adjuvant to phototherapy in neonates with hyperbilirubinemia is associated with significant reduction of serum bilirubin levels. (Khafaga et al., 2022) The present study is to compare the effects of Fenofibrate adjuvant to phototherapy with conventional phototherapy for exaggerated neonatal hyperbilirubinemia in the form of bilirubin reduction, duration of phototherapy, hospital stay & observation of side-effects.

Administration of a single dose of fenofibrate as an adjunct along with phototherapy to neonates showed a significant reduction of serum bilirubin and duration of phototherapy. The duration was shorter in the fenofibrate group in comparison to the control group. No side effects of fenofibrate were observed after a single dose administration. (Islam et al., 2021) Newborns admitted in neonatal units of pediatric medicine unit I, Services Hospital Lahore and fulfilling the inclusion & exclusion criteria will be the study subject. The patients will be divided randomly into two groups i.e., group A (intervention) and group B (non-intervention). Randomization will be performed by using computer generated numbers.

The parent/guardian of the neonate will be informed about the study verbally and informed consent will be taken. The demographic data will be obtained, detailed history regarding symptoms, onset of disease, duration of illness, progression and medication will be taken. General physical examination and systemic examination will be carried out.

In babies with jaundice, clothes will be taken off but eyes and genitalia will be covered. Baby will be kept under phototherapy at baby-to-light distance of 20-40 cm (Gomella, ed. 2013) with changing position every 2 hourly to expose as much part as possible. Single dose of Fenofibrate will be given to the group A (intervention group) at dose of 10mg/Kg (Al-Asy et al., 2015). Group B (non-intervention) will only be given phototherapy. Then every 24-hourly sample for serum bilirubin will be sent for lab analysis, for 3 days. Fenofibrate is readily available in market as 200mg & 67mg generic capsule which will be diluted with sterile distilled water in syringe dropper & calculated amount of dose will be given orally.

Outcome of this study will be measured by number of days needed for serum bilirubin to decrease below phototherapy range in both groups. If the role of Fenofibrate is established in the management of exaggerated physiological hyperbilirubinemia in newborns, it will be beneficial to minimize the risk of the complications off prolong phototherapy.

ELIGIBILITY:
Inclusion Criteria:

* Newborn of either sex of age 2nd day of life to 14th day of life.
* Exaggerated physiological jaundice without identifiable cause.
* Full-term newborn ≥37 to ≤42 weeks of gestation with birth weight >2.5kg
* Total serum bilirubin level within phototherapy range (NICE Guidelines)

Exclusion Criteria:

* Preterm newborn < 37 weeks of gestation or low birth weight <2.5kg
* Direct hyperbilirubinemia (Conjugated Bilirubin >2mg/dl or >10% of Total Serum Bilirubin)
* Pathological jaundice due to lab proven Sepsis / Blood Group Incompatibility.

Ages: 24 Hours to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 156 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
number of days needed for serum bilirubin to decrease below phototherapy range | 72 hours
  number of days needed for serum bilirubin to decrease below phototherapy range in both groups

SECONDARY OUTCOMES:
Hospital length of Stay | 72 hours
  number of days

CONTACTS AND LOCATIONS:
Overall Officials: Tayyaba K Butt, FCPS, MRCPCH, Study Chair — Professor & Head of Department of Pediatrics
Locations (1):
- Services Institute of Medical Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR) Analytic Code
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year
Access Criteria: open

REFERENCES:
- [Background] Awad MH, Amer S, Hafez M, Nour I, Shabaan A. "Fenofibrate as an adjuvant to phototherapy in pathological unconjugated hyperbilirubinemia in neonates: a randomized control trial.". J Perinatol. 2021 Apr;41(4):865-872. doi: 10.1038/s41372-020-00861-2. Epub 2020 Oct 17. PMID 33070152